CLINICAL TRIAL: NCT00812539
Title: A Randomized Clinical Trial of a Secure Website Shared Between Patients and Providers for Blood Glucose Monitoring in Type-2 Diabetes
Brief Title: Diabetes Connect: Patients and Providers Use of a Secure Website for Blood Glucose Monitoring in Type-2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Director, Center for Connected Health, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2008-P-001898/1; MGH
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Blood glucose monitoring; Internet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetes Connected Health Tool "Deluxe" (Experimental): Subjects enrolled into the intervention arm will measure their glucose levels by using a glucometer. An iMetrikus modem will upload the blood glucose readings to a secure, web-based portal. Participants will be given login information to access this portal, where they can view their glucose readings and detailed graphical representation of their blood glucose levels over time, read educational material regarding diabetes management and receive personalized tips and feedback from their physicians (who will also have access to these subjects' information on the web portal).
  Interventions: Other: Subject/Provider Portal "Diabetes Connected Health" tool - Deluxe
- Diabetes Connected Health Tool "Basic" (Active Comparator): Control group will measure their glucose levels by using a glucometer. An iMetrikus modem will upload the blood glucose readings to a secure, web-based portal. Participants will be given login information to access this portal. where they can view their glucose readings in tabular form. Their physicians will not have access to this information.
  Interventions: Other: Subject only Portal "Diabetes Connected Health Tool" Basic

INTERVENTIONS:
Other: Subject/Provider Portal "Diabetes Connected Health" tool - Deluxe — Subjects enrolled into the "Deluxe"intervention will use a glucometer, a modem to upload the blood glucose readings to a secure, web-based portal ("Diabetes Connected Health" tool) where they can view detailed graphical representation of their blood glucose levels over time, educational material regarding diabetes management and receive personalized tips and feedback from their physicians (who will also have access to their subjects' information on the web portal and contact them by an embedded messaging system). Subjects with new high or low readings will be flagged. Providers can initiate messages to subjects regarding symptoms or medications. A medication summary and log of all readings uploaded with date/time will be displayed on the website as well as a graphical display of all uploaded glucose readings over time and will allow subjects to enter comments regarding each critical reading.
  Arms: Diabetes Connected Health Tool "Deluxe"
Other: Subject only Portal "Diabetes Connected Health Tool" Basic — Patients enrolled in the Diabetes Connect "Basic" intervention will use a glucometer, a modem which will upload the blood glucose readings to a secure, web-based portal (the "Diabetes Connected Health" tool) where they can view their readings in a less detailed/journal fashion. No detailed graphical representation of their blood glucose levels over time is available to this group, nor is any educational material regarding diabetes management. Their physicians will not have access to these subjects' information on the web portal and will not have the ability to contact them by an embedded messaging system.
  Arms: Diabetes Connected Health Tool "Basic"

SUMMARY:
Currently, diabetic patients who receive their care at the diabetes clinic self monitor their blood glucose using a portable glucometer, under the direction of care providers at the clinic. We propose to conduct a randomized controlled trial to examine the effect of the "Diabetes Connected Health" tool, which is a secure website shared between patients of Type-2 Diabetes and their providers and displays (subjects') blood glucose values in graphical format. The study will be carried out through multiple primary care practices within the Partners/PCHI Network. We hypothesize that implementation of the Diabetes Connected Health Tool will result in overall better Diabetes Care, in terms of improved patient-provider interaction, and better patient satisfaction towards their care.

DETAILED DESCRIPTION:
The study will be carried out at multiple practices within Partners HealthCare system and will have one Intervention and one control arm.

Subjects enrolled into the intervention arm will use a OneTouch Ultra2 glucometer and an iMetrikus modem device which will upload the blood glucose readings to a secure, login-enabled web-based portal. Subjects will be given login information to access to their own individual Internet site, where they can view their readings and detailed graphical representation of their blood glucose levels over time, read educational material regarding diabetes management and receive personalized tips and feedback from their physicians (who will also have access to their patients' information on the web portal).

Subjects enrolled into the control arm will have access to the same glucometer and modem, and will have access to another individual internet website (the "Basic Site") which will show their glucose readings and graphical representation of glucose levels. Each patient will be enrolled for 3 months. and the primary outcome measure will patient and provider satisfaction with the Diabetes Connected Health tool.The specific aims along with hypothesis of the study are:

1. To develop a web-based application ("Diabetes Connected Health") that will enable home-based glucose monitoring results to be readily incorporated into clinical glycemic management.

   Hypothesis: We hypothesize that through a development process incorporating interactive feedback loops between software developers, patients, clinicians, and other stakeholders, we can create a web-based clinical application that will be adopted by clinical practices.
2. To test the impact of the "Diabetes Connected Health" tool in a randomized clinical trial.

Hypothesis: We hypothesize that implementation of the tool will have a beneficial impact relative to control patients in several critical domains:

Patient Domains

1. Increase patients' knowledge of their diabetes management plan.
2. Increase patients' satisfaction with their clinical care.
3. Increase patients' awareness of why they have high and/or low glucose readings.
4. Increase patients' satisfaction with patient-provider communication.

Provider Domains

1. Increase clinician satisfaction with clinical care.
2. Increase clinician knowledge of individual patient care issues.

ELIGIBILITY:
Eligibility Criteria for Partners HealthCare practices:

Manage type-2 Diabetes patients.

Have at least one non-Physician provider (nurse practitioner, nurse, diabetes educator) with responsibility for diabetes patient care

Inclusion Criteria for subject selection:

Diagnosis of type 2 diabetes

Age 18 years or older

English speaking/able to read English

Last measured Hemoglobin A1c (HbA1c) > 7.5 % in the last 12 months.

Prescribed glucose self-monitoring, and either currently self monitoring or willing to monitor their blood glucose, as prescribed by their care provider, using the OneTouch Ultra2 portable glucometer.

Access to the Internet for the 6 months the study will run.

Access to a compatible analog telephone line at either their work place or home such that the subjects are able to upload the glucometer readings to the website.

Access to an active email account.

Receiving diabetes care primarily within the practice.

Exclusion Criteria for subject selection:

Subjects having mental health, cognitive or physical impairments that would preclude the set up and use of the modem, glucometer or computer.

Subjects are not candidates for guideline-based diabetes care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Subject and provider satisfaction with the intervention. | Upon completion of the trial.

SECONDARY OUTCOMES:
Subject knowledge of diabetes and motivation | On completion of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Richard W. Grant, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Partners HealthCare Hospitals/Clinics (Massachusetts General Hospital, Brigham and Womens Hospital), Boston, Massachusetts, United States